CLINICAL TRIAL: NCT04396951
Title: Clinical Optimization of Ambient Temperature and Heating Methods in Caring in Major Burns Patients
Brief Title: Optimal Heating Temperature in Major Burns Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: University of Valladolid (Other); Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Alonso Fernández, Juan Manuel, Master of Science in Nursing, University Rovira i Virgili
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HEATINGBURNS01
Record Dates: First submitted 2020-05-06; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Burns; Thermal Injury; Nurse's Role
Keywords: Nursing; energy metabolism; hypothermia; heating; burns; thermoregulation
MeSH Terms: conditions — Burns; Hypothermia

STUDY DESIGN:
Intervention Model Description: A pre and post intervention quasi-experimental epidemiological study without control group, will be carried out in large burned patients that will assess the influence on the metabolic expenditure of the inclusion of active external reheating in the control of the environmental temperature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive external overheating (No Intervention): Passive external overheating in the environmental temperature control adjusted to thermal comfort.
  Measure during 6 hours with indirect calorimetry
- Active external overheating with heating plate (Active Comparator): Combination of passive and active external heating with heating plate Measure during 6 hours with indirect calorimetry
  Interventions: Device: Active external overheating with heating plate, Aragonia ® MTC 400
- Active external overheating with air blanket (Active Comparator): Combination of passive and active external heating with convective air blanket Measure during 6 hours with indirect calorimetry
  Interventions: Device: Active external overheating with air blanket, Equator Level 1® de Smiths Medical

INTERVENTIONS:
Device: Active external overheating with heating plate, Aragonia ® MTC 400 — It is a heating device that is adjustable in height up to 50 cm from the patient and generates radiant heat at low temperature (up to 39 ◦C) distributed evenly. It is equipped with an adjustable 0-9 potentiometer and has a skin temperature probe as a control and safety mechanism Measure during 6 hours with indirect calorimetry in first week
  Other Names: Aspira Medical AB Aragonia ® MTC 400. Certificate CE 0413
  Arms: Active external overheating with heating plate
Device: Active external overheating with air blanket, Equator Level 1® de Smiths Medical — Composed of a unit that produces hot air and forced air adjustable from 38ºC to 43ºC. Sends hot forced air distributed by tubular blanket that convectively heats the patient by diffusing hot air directed at the patient through the textile pore of the air blanket Measure during 6 hours with indirect calorimetry in first week
  Other Names: Equator Level 1® de Smiths Medical REF EQ-5000. Certificate CE 0473
  Arms: Active external overheating with air blanket

SUMMARY:
pre and post intervention quasi-experimental epidemiological study without a control group will be carried out in large burned patients that will evaluate the influence on metabolic expenditure of the inclusion of active external rewarming in the control of body temperature.

DETAILED DESCRIPTION:
the heavily burned patient requires specific care to prevent hypothermia and maintain body temperature. You are at high risk of developing hypothermia in the acute phase due to heat losses from convection, radiation, evaporation, and conduction. After the acute phase, the patient due to physiological mechanisms and the hypermetabolic response mainly demands a temperature close to 38.5ºC, ruling out the infectious focus. According to the authors, environmental temperatures between 28-33ºC are recommended for the care of these patients to decrease energy expenditure. The research carried out has studied the influence of passive external heating (environmental regulation), without including the influence of active external heating (heat blankets, heating plate ...) or the study of the thermal comfort of large burned patients and of professionals who provide them they attend.

A pre and post intervention quasi-experimental epidemiological study without a control group will be carried out in large burned patients that will evaluate the influence on metabolic expenditure of the inclusion of active external rewarming in the control of body temperature. Metabolic expenditure will be measured by indirect calorimetry in the usual treatment with passive external rewarming and post-intervention in the combination of passive and active external heating. The combination of passive and active external reheating will previously study the operating temperature in various cases for optimal application, as well as the definition of thermal comfort in the large burn unit. The specific training of the personnel involved in the care of these patients will be required for the application of the evidence-based recommendations and the evaluation of their implementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with thermal burns.
* Patient with high burn criteria according to ABA:
* 2nd degree burn
* Patient 18 - 59 years: SCQ> 20%
* Patient> 60 years or pathology: SCQ> 10%
* 3rd degree burn
* SCQ> 10%
* Patients on mechanical ventilation

Exclusion Criteria:

* Sepsis criteria according to ABA.
* Enzyme debridement application (data within 24 hours).
* 6 hours after a surgical intervention.
* After 2 hours after healing burns
* Patients in hemorrhagic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic expenditure | Measure during 6 hours with indirect calorimetry in first recovery week with three heating methods
  Compare the metabolic expenditure of burned patients according to the heating method between the combination of active and passive external adjusted to thermal comfort versus external passive overheating.

SECONDARY OUTCOMES:
Optimal environmental temperature | Measure during 6 hours with three heating methods in first recovery week
  Define the optimal environmental temperature according to the characteristics of the patient with a large burn during the acute phase, assigning the available resources.
Thermal comfort | Measure during 6 hours with three heating methods first recovery week
  Analyze thermal comfort according to heating methods in large burned patients.

OTHER OUTCOMES:
Nursing care planning | Measure Scales during three heating methods in six hours, first recovery week
  Evaluate the nursing care plan in the thermoregulation of the burned patient according to the standardized nurse taxonomy.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Alonso Fernández, MSN, Principal Investigator — Sanidad Castilla y León

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT04396951/Prot_SAP_ICF_000.pdf